CLINICAL TRIAL: NCT02384044
Title: A Pilot Clinical Study to Evaluate the Safety and Efficacy of Marketed Oxalate Strips Compared to a Marketed Safety Pen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015012
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

ARMS (2):
- Crest® Sensi-Stop™ Strips (Active Comparator): Professionally Applied
  Interventions: Device: Crest® Sensi-Stop™ Strips
- Colgate® Sensitivity Relief Pen (Active Comparator): Professionally Applied
  Interventions: Device: Colgate® Sensitivity Relief Pen

INTERVENTIONS:
Device: Crest® Sensi-Stop™ Strips
  Arms: Crest® Sensi-Stop™ Strips
Device: Colgate® Sensitivity Relief Pen
  Arms: Colgate® Sensitivity Relief Pen

SUMMARY:
This pilot study will evaluate the safety and effectiveness of a marketed sensitivity strip on existing dentinal hypersensitivity compared to a marketed sensitivity pen.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* sign an informed consent form and be given a copy
* be in good general health as determined by the Investigator/designee
* agree to delay any elective dentistry, including dental prophylaxis, and to report any dentistry received during the course of the study
* agree to not participate in any other oral care study for the duration of this study
* agree to return for scheduled visits and follow all study procedures
* have dentinal hypersensitivity with at least one tooth with a Schiff sensitivity score of at least 1 in response to the cold water challenge

Exclusion Criteria:

* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession
* active treatment for periodontitis
* any diseases or conditions that might interfere with the subject safely completing the study
* inability to undergo study procedures
* fixed facial orthodontic appliances
* a history of kidney stones
* self-reported pregnancy or nursing
* known allergies to the following ingredients; aqua, glycerin, cellulose gum, dipotassium oxalate, carbomer, sodium hydroxide, sodium benzoate, and potassium sorbate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Gerlach, DDS, MPH, Principal Investigator — Procter and Gamble
Locations (1):
- Oral Health Science Center, Mason, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crest® Sensi-Stop™ Strips: Professionally Applied
  Crest® Sensi-Stop™ Strips
- Colgate® Sensitivity Relief Pen: Professionally Applied
  Colgate® Sensitivity Relief Pen
Period: Overall Study
Arm/Group | Crest® Sensi-Stop™ Strips | Colgate® Sensitivity Relief Pen
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crest® Sensi-Stop™ Strips | Colgate® Sensitivity Relief Pen | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (7.97) | 43.5 (7.77) | 43.4 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 9 | 5 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Oriental | 0 | 1 | 1
  Black | 1 | 1 | 2
  Caucasian | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Visual Analog Scale
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced. A negative change from Baseline score represents a decrease in sensitivity from baseline.
Time Frame: 1 Day
Population: Thirty (30) subjects received study products and completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips | Colgate® Sensitivity Relief Pen
Number analyzed (Participants) | 15 | 15
Units on a scale | -22.933 (19.252) | -3.200 (11.857)

2. Secondary Outcome: Change From Baseline for Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A negative change from Baseline score represents a decrease in sensitivity from baseline.The mean change from Baseline was calculated for this measure.
Time Frame: 1 Day
Population: Thirty (30) subjects received study product and completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips | Colgate® Sensitivity Relief Pen
Number analyzed (Participants) | 15 | 15
Units on a scale | -0.800 (0.561) | 0.000 (0.378)

ADVERSE EVENTS:
Arm/Group | Crest® Sensi-Stop™ Strips | Colgate® Sensitivity Relief Pen
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crest® Sensi-Stop™ Strips (N=15) | Colgate® Sensitivity Relief Pen (N=15)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cheilitis
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes